CLINICAL TRIAL: NCT01132235
Title: An Open-label Study to Evaluate the Efficacy of Re-treatment for Patients With a History of Etanercept Use
Acronym: ENBRECAP2009
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Florida Academic Dermatology Centers (Other)
Collaborators: Amgen (Industry)
Responsible Party: Francisco A Kerdel, M.D., Florida Academic Dermatology Centers
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENBRECAP2009
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: etanercept — 50mgs subcutaneous injections twice a week for 12 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy of re-treatment with etanercept 50mg subcutaneous injections twice weekly for 12 weeks in subjects who have previously been treated etanercept and efficacy diminished.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with psoriasis who have previously been treated with etanercept for a minimum of 6 months and discontinued treatment due to loss of efficacy. Every attempt will be made to obtain loss of efficacy history from the subject's medical chart;when etanercept was commenced and terminated and description of patient's psoriasis on termination and details of new treatment commenced. Subjects must have failed their latest psoriasis treatment after a period of three months. This will be measured as a PGA of ≥ 3.
* There is no specific requirement as to when prior treatment with etanercept occurred and no requirement as to what type of treatment(s) used between initial and subsequent treatments.
* Are ≥ 18 years of age
* PGA ≥ 3
* BSA minimum of 5%

Tuberculosis inclusion criteria

* Have no history of latent or active TB prior to screening.
* Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination.
* Have had no recent close contact with a person with active TB.
* Within 1 month prior to the first administration of study have a negative tuberculin skin test.

  * The ability to give written informed consent and comply with study procedures.

Exclusion Criteria:

* Current enrollment in any other investigational device or investigational drug trial(s), or receipt of any other investigational agent(s) within 28 days before baseline visit.
* Known hypersensitivity to Enbrel® (etanercept) or any of its components or known to have antibodies to etanercept.
* Latex sensitivity [NB: only applicable if they are using prefilled syringe or prefilled SureClick™ autoinjector presentations]
* Prior or concurrent use of cyclophosphamide therapy
* Concurrent sulfasalazine therapy.
* A positive HBV test or known history of any other immuno-suppressing disease.
* Any mycobacterial disease or high risk factors for tuberculosis (TB), such as family member with TB, positive purified protein derivative (PPD) or taking anti-tuberculosis medication.
* Active or chronic infection within 4 weeks before screening visit, or between the screening and baseline visits.
* History of listeriosis, histoplasmosis, chronic or active Hepatitis B infection and Hepatitis C, human immunodeficiency virus (HIV) infection, immunodeficiency syndrome, chronic recurring infections or active TB, or other opportunistic infections
* If etanercept was previously discontinued due to a serious adverse event
* Severe comorbidities (diabetes mellitus requiring insulin; CHF of any severity; or myocardial infarction, cerebrovascular accident or transient ischemic attack within 6 months of screening visit; unstable angina pectoris; uncontrolled hypertension (sitting systolic BP <80 mm Hg or > 160 or diastolic BP > 100 mm Hg); oxygen-dependent severe pulmonary disease; history of cancer within 5 years [other than resected cutaneous basal or squamous cell carcinoma of the skin or in situ cervical cancer])
* Systemic lupus erythematosus, history of multiple sclerosis, transverse myelitis, optic neuritis or seizure disorder.
* Use of a live vaccine 90 days prior to screening visit, or concurrent use of a live vaccine.
* Any condition or circumstances judged by the patient's physician [or the investigator or medically qualified study staff] to render this clinical trial detrimental or otherwise unsuitable for the patient's participation.
* Female subjects who are pregnant, nursing or planning pregnancy (both men and women) and not using acceptable methods of birth control during the trial (hormonal, barriers, abstinence).
* Women who are breast feeding

History of non-compliance with other therapies.

* History of alcohol abuse within the last 12 months
* Concurrent use of anakinra
* Subjects who cannot discontinue any of the drugs below for 2 weeks prior to the baseline visit or during the study;

A two week wash out period is appropriate as it would be unethical to expect subjects whose disease if flaring to remain untreated for a longer period of time. The first dose of etanercept will be administered two weeks after the last biologic dose.

* Immunosuppressants, antimalarials, or sulfasalazine.
* Other Ani-TNFs
* Cyclosporine
* Efalizumab
* Azathioprine
* Hydroxyurea
* Live vaccines
* Tacrolimus
* Oral retinoids (isotretinoin,acitretin,bexarotene)
* Ultra violet light therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving a Physician's Global Assessment (PGA) score of minimal (1) or clear (0) at week 12. | 12 weeks
  Physician's Global Assessment (PGA) score of minimal (1) or clear (0) at week 12 will measure efficacy of retreatment with etanercept

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Academic Dermatology Center, Miami, Florida, United States